CLINICAL TRIAL: NCT05333770
Title: Repetitive Transcranial Magnetic Stimulation as a Means to Promote CST Axon Regeneration in Persons With Spinal Cord Injury
Brief Title: Repetitive Transcranial Magnetic Stimulation to Promote Regeneration in Persons With SCI
Acronym: rTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-1107-20
Record Dates: First submitted 2021-10-11; First posted 2022-04-19 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SCI Group (Experimental): Complete testing at Baseline, Post, and 6 month follow up. Intervention includes 15 treatment sessions (3-5 times per week) with HF-rTMS & 6 month follow-up. Following HF-rTMS, there will be 30 minutes of arm and hand training. Each session will last for approximately 60 mins.
  At baseline, post and 6 months, the following evaluations to evaluate safety and other related measures. These measures include a safety and pain questionnaire, spasticity measurement, a physician or clinician evaluation to determine motor and sensory neurological level of injury, hand and arm function measurement, evaluation of ability to perform everyday tasks, and measures to determine level of brain function.
  Interventions: Device: High-frequency repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: High-frequency repetitive transcranial magnetic stimulation — TMS is an investigational device that provides a way to test the function of a specific part of the brain that is devoted to moving my affected upper limbs by directing a low electrical current to that part of the brain through the scalp.

SUMMARY:
This is a research study to evaluate the safety, efficacy and feasibility of high-frequency repetitive transcranial magnetic stimulation (HF-rTMS) in patients with subacute spinal cord injury.

DETAILED DESCRIPTION:
This research study is investigating whether repetitive high-frequency transcranial magnetic stimulation (HF-rTMS) in patients with subacute spinal cord injury is safe, efficacious, and feasible. The study will take approximately 7-8 months to complete, during which 15 training sessions with HF-rTMS will be completed. Followed by 30 minutes each session of arm and hand training without HF-rTMS. The participants will complete testing after the 15 training sessions as well as 6 months following completion.

ELIGIBILITY:
Inclusion Criteria:

* Be less than 8 weeks post injury
* Must have an incomplete spinal cord injury at a neurological level of injury between the C2-C6 level and an impairment grade A, B, C, or D, according to the American Spinal Injury association (ASIA) Impairment Scale
* If an outpatient, will be at least 6 months post injury

Exclusion Criteria:

* Have a pacemaker
* Have metal in the skull
* Have a history of seizures, or a brain injury
* Being pregnant
* Have skin issues or open wounds
* Have severe contractures and/or spasms in my elbow/wrists as determined by study staff examination at screening
* Study staff will review medications to determine if taking any drugs that would increase risk of having a seizure while undergoing TMS. If taking such medications, will not be enrolled

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Neuro Recovery Scale (NRS). | 6 months
  Measure of the degree a person who has sustained a spinal cord injury (SCI) has recovered the ability to perform functional tasks relative to how the individual performed these tasks prior to injury. The NRS consists of a numeric version of the visual analog scale. The most common form of the NRS is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible. This type of scale can be administered verbally.
GRASSP | 6 months
  The Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) is an extensive and validated impairment and functional measure which is able to detect subtle neurologic changes in individuals with spinal cord injury.
  Specifically, it evaluates the domains of sensation, strength, quality of different grip patterns and the ability to complete a variety of functional tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No